CLINICAL TRIAL: NCT00174824
Title: Evaluation of Diabetic Retinopathy Progression in Subjects With Type 2 Diabetes Mellitus Treated With Insulin
Brief Title: Comparison of Insulin Glargine and NPH Human Insulin in Progression of Diabetic Retinopathy in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTS6036
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Diabetic Retinopathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Diabetic Retinopathy | interventions — Insulin Glargine

INTERVENTIONS:
Drug: Insulin glargine

SUMMARY:
To compare the progression of diabetic retinopathy in type 2 diabetic patients with mild-to-moderate diabetic retinopathy treated with insulin glargine vs NPH human insulin.

DETAILED DESCRIPTION:
Randomized, open-label assignment of type 2 patients who are on a stable antidiabetic regimen to treatment with either insulin glargine or BID NPH human insulin, with baseline diabetic retinopathy of severity 53/<53 on the ETDRS scale, for 5 years of followup. Outcomes measured by seven-field fundus photography at baseline, 1.5, 3,6,and 9 months, and annually.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus for at least 1 year
* treated with oral antidiabetic agents or insulin at stable doses for at least 3 months
* HbA1c between 6 and 12% inclusive
* baseline retinopathy severity not to exceed 53/<53 on the ETDRS scale
* unlikely to require laser surgery or vitrectomy within upcoming year

Exclusion Criteria:

* prior treatment with insulin glargine
* treatment with insulin analogs (eg insulin lispro or aspart) in the year prior to enrollment

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1024 (Actual)
Dates: Start 2001-06; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with a 3-step or greater progression in the patient
level recoded integer ETDRS retinopathy scale

SECONDARY OUTCOMES:
The percentage of patients who:develop proliferative retinopathy or develop clinically significant macular edema
the distribution of patients on the patient level recoded integer ETDRS retiopathy scale
the change from baseline in HbA1c and fasting plasma glucose
the incidence of hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (2):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Laval, Canada

REFERENCES:
- [Derived] Semlitsch T, Engler J, Siebenhofer A, Jeitler K, Berghold A, Horvath K. (Ultra-)long-acting insulin analogues versus NPH insulin (human isophane insulin) for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD005613. doi: 10.1002/14651858.CD005613.pub4. PMID 33166419
- [Derived] Rosenstock J, Fonseca V, McGill JB, Riddle M, Halle JP, Hramiak I, Johnston P, Davis M. Similar progression of diabetic retinopathy with insulin glargine and neutral protamine Hagedorn (NPH) insulin in patients with type 2 diabetes: a long-term, randomised, open-label study. Diabetologia. 2009 Sep;52(9):1778-88. doi: 10.1007/s00125-009-1415-7. Epub 2009 Jun 13. PMID 19526210